CLINICAL TRIAL: NCT03201029
Title: Assessment of Dermatologists at Skin of Color Clinics
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Principal Investigator, Northwestern University
Other Study IDs: SP02072017
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Characteristics of Dermatologists Who Focus on Ethnic Skin
Keywords: center for ethnic skin; skin of color clinic; ethnic skin center

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As a physician, narrowing ones' practice to a particular pathology or group of people is common. Dermatologists are able to concentrate within a number of different areas: cancer, cosmetics, pediatrics or ethnic populations to name a few. Recently, there has been an emphasis on developing skin of color (SOC) clinics and recruiting dermatologists who focus on skin diseases that effect patients with skin of color. In this study, patients with SOC is defined to encompass that of persons of African, Asian, Native American, Middle Eastern, and Hispanic backgrounds. An emphasis on SOC benefits patients in a variety of ways: 1) these dermatologists are trained to recognize pathology that may present differently, depending on the Fitzpatrick skin type and ethnicity of the patient, 2) these dermatologists are trained to address medical disparities that are present among patients with SOC, 3) these dermatologists are trained to address culturally sensitive topics that may be common among patients with SOC. Despite the growing number of SOC patients and the benefit that SOC clinics provide, studies have not looked at the characteristics that influence dermatologists to focus on SOC as opposed to other specialty areas. Therefore, we aim to identify information that may influence dermatologists to focus on skin disease prevalent among patients with SOC.

Currently, there are nine academic institutions with an Ethnic Skin Center in the United States. Given the limited number of academic centers with a designated center focused on SOC, a lot of care of skin of color patients happens in private practices. This is supported by the fact that many of the members in the Skin of Color Society are dermatologists in private practices. Thus, SOC clinic is defined broadly in our study to encompass not only academic dermatologists but also private practice dermatologists who have special interest in care of skin of color patients. Regardless of the type of practice, we hope to identify unique characteristics of dermatologists focusing on SOC skin diseases.

DETAILED DESCRIPTION:
Dermatologists who are members of the Skin of Color Society practicing in the US will be sent a recruitment letter in the mail that includes a description of the study and paper survey. The survey will collect participant first and last name so the research team can track replies. Participant first and last name will not be transferred from the surveys and not used in data analysis. Even though it is likely that there are dermatologists with practices involving skin of color patients or with interest in skin of color patients who are not members of the Skin of Color Society, we believe that this will be a representative group of physicians with this interest. We do not believe we will experience significant bias. Duration of the subjects' involvement will be approximately 10 minutes. The total participant recruitment period will be approximately 8 weeks. Quantitative survey responses will be compiled, coded, and entered into a statistical program.

ELIGIBILITY:
Inclusion Criteria:

* Dermatologists at known SOC clinics (both academic and private) practicing in the United States who are members of the Skin of Color Society.
* Dermatologists who identify skin of color patients as an area of interest.

Exclusion Criteria:

* Subjects who do not speak English.
* Subjects without a mailing address.
* Dermatologists who are not members of the Skin of Color Society.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: dermatologists at skin of color clinics
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Demographic Characteristics | 2 months
  Gender, ethnicity, name of the institution of training, and zip code of the location of practice will be collected through a paper survey and statistically analyzed. The unit of measure would be the number of survey participants.
Method of learning | 2 months
  Method of learning about skin diseases prevalent in skin of color patients of dermatologists who focus on patients with skin of color will be collected through a paper survey and will be statistically analyzed. The unit of measure would be the number of survey participants.

CONTACTS AND LOCATIONS:
Overall Officials: Stavonnie Patterson, MD, Principal Investigator — Northwestern University; Roopal Kundu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor SC. Skin of color: biology, structure, function, and implications for dermatologic disease. J Am Acad Dermatol. 2002 Feb;46(2 Suppl Understanding):S41-62. doi: 10.1067/mjd.2002.120790. PMID 11807469
- [Background] Kundu RV, Patterson S. Dermatologic conditions in skin of color: part I. Special considerations for common skin disorders. Am Fam Physician. 2013 Jun 15;87(12):850-6. PMID 23939567
- See also: Skin of Color Society website — http://skinofcolorsociety.org/